CLINICAL TRIAL: NCT00992004
Title: Comparative, Randomized, Double-blind, Placebo-controlled, Parallel Group Study, to Evaluate the Efficacy of a Turmeric Extract (Arantal®) Versus Placebo in Patients With Osteoarthritis of the Knee (Gonarthrosis).
Brief Title: Evaluation of the Efficacy of a Turmeric Extract (Arantal®) in Patients With Osteoarthritis of the Knee (Gonarthrosis).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bioxtract SA (Industry)
Collaborators: Nukleus (Industry)
Responsible Party: Dr Ingrid Jacquemond-Collet, bioXtract SA
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARKOS; 2009-A00174-53
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2010-05

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, Knee; Osteoarthritis; Joint Diseases; Arthritis; Rheumatic Diseases
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Joint Diseases; Arthritis; Rheumatic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arantal® (Experimental): Highly bioavailable turmeric extract (food supplement)
  Interventions: Dietary Supplement: Arantal® (highly bioavailable turmeric extract)
- Placebo (Placebo Comparator): Same capsule without the active ingredients (only excipients)
  Interventions: Dietary Supplement: Arantal® (highly bioavailable turmeric extract)

INTERVENTIONS:
Dietary Supplement: Arantal® (highly bioavailable turmeric extract) — 4 capsules a day, before breakfast

SUMMARY:
The purpose of this study is to determine the efficacy and the tolerance on 15 days of a turmeric extract (Arantal®) on pain related to gonarthrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 40 through 80 years of age
* Subject diagnosed with femorotibial osteoarthritis of the knee (diagnosed according to the clinical and radiologic criteria of ACR),
* Patient's Assessment of Arthritis Pain measurement on the last 24 hours of at least 50 mm on VAS,
* Patient has not received any NSAIDs within 72 hours and any analgesics within 24 hours,
* Patients with chronic knee pain (i.e., knee pain at least every other day during the month preceding inclusion),
* Patients with radiologic knee osteoarthritis (Kellgren-Lawrence grade 2-4, on radiography less than 12 months old),
* Patients having signed the informed consent,
* Patients capable of comprehend the study instructions.

Exclusion Criteria:

* Related to the osteoarthritis pathology:

  * Osteoarthritis linked to a metabolic arthropathy: chondrocalcinosis already diagnosed or defined by calcium edging on at least one femorotibial joint space, gout...,
  * Predominant associated symptomatic femoropatellar osteoarthritis,
  * Chondromatosis or villonodular synovitis of the knee,
  * Recent trauma (< 1 month) of the knee responsible for the pain,
  * Knee joint effusion justifying an evacuation through puncturing,
  * Inflammatory flare (night pain, joint effusion) corresponding to a KOFUS score less than 7,
  * Pathology potentially interfering with the evaluation (metabolic inflammatory arthropathy, rheumatoid arthritis, lower limb radiculalgia, arthritis...),
* Related to previous and associated treatments:

  * Corticosteroids injection in the previous month, whatever the joint concerned,
  * Hyaluronan injection in the evaluated knee during the previous 6 months,
  * Patient who took NSAID in the 72 hours prior to inclusion or Analgesics in the 24 hours prior to inclusion,
  * Slow-acting drugs for OA and/or dietary supplements taken within less than 3 months prior to the study product administration or for which the dose has been modified in the last three months (ex: chondroitin sulfate, diacerein, soy and avocado unsaponifiables, oxaceprol, granions de cuivre, glucosamine, phytotherapy for OA, homeopathy for OA...),
  * Anticoagulant treatment without gastric protection,
  * General corticotherapy,
  * Contraindication to paracetamol.
* Related to associated pathologies:

  * Patient suffering from serious associated illness (liver failure, kidney failure, non-controlled cardiovascular diseases...),
  * Peptic ulcer.
* Related to patients:

  * Pregnant or breastfeeding women
  * Pre-menopausal women with no contraception
  * Patients unable to write
  * Patients enrolled in a clinical trial in the previous 3 months
  * Patients under juristic protection or under guardianship.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Patient's Assessment of Arthritis Pain using a Visual Analogue Scale (OA-Pain VAS) | 15 days

SECONDARY OUTCOMES:
Kinetics of the analgesic effect by a variance analysis in repeated measures (Likert Scale) | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Yves Henrotin, Pr, Principal Investigator — University of Liege - Bone and Cartilage Research Unit
Locations (1):
- Henri Mondor Hospital, Créteil, France